CLINICAL TRIAL: NCT04687657
Title: Application of Umbilical Cord Blood Transfusion in Consolidation Therapy of Elderly Patients With Acute Myeloid Leukemia
Brief Title: Umbilical Cord Blood Transfusion in Consolidation Therapy of Elderly Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-016
Record Dates: First submitted 2020-12-27; First posted 2020-12-29 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Myelomonocytic, Acute
Keywords: Leukemia, Myelomonocytic, Acute; Umbilical cord blood transfusion; treatment effect
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cord blood transfusion (Experimental): The arm that will receive the target treatment.
  Interventions: Drug: umbilical cord blood

INTERVENTIONS:
Drug: umbilical cord blood — During the consolidation chemotherapy stage, the umbilical cord blood transfusion is given twice (interval of 1 month) to support treatment. On the first day after umbilical cord blood transfusion, the proportion of NK cells in peripheral blood is detected. If it is less than 20%, the NK cells sre activated by subcutaneous injection of recombinant human interleukin-2 (rhIL-2) on the second day after infusion.
  Other Names: cord blood

SUMMARY:
After complete remission, elderly AML patients cannot tolerate hematopoietic stem cell transplantation and standard-dose consolidation chemotherapy, and the 5-year survival rate is around 10%. Therefore, it is necessary to explore treatment strategy that can support chemotherapy or improve immunity. Umbilical cord blood is rich in hematopoietic stem cells and immune cells. However,Cord blood transplantation for adults is still being explored. The application of cord blood in supportive treatment can be actively explored. Cord blood has low immunogenicity and is unlikely to cause Graft versus host disease (GVHD), and the infusion is relatively safe. The Department of Hematology of Shanghai Ruijin Hospital has conducted a related phase II clinical study, and found that cord blood transfusion reduced the chance of infection and increased the 2-year survival. Our subject is a prospective single-arm clinical study. It is planned to recruit 20 elderly AML patients to explore whether the application of cord blood infusion can further improve the prognosis of patients during their consolidation chemotherapy.

DETAILED DESCRIPTION:
20 elderly AML patients who achieved complete remission (CR) after induction chemotherapy will be enrolled in this study. Baseline data are collected and informed consents are signed before consolidation chemotherapy. At the same time, HLA typing test is carried out, and the corresponding cord blood is matched from the cord blood bank. During the consolidation chemotherapy stage, the cord blood transfusion is given twice (interval of 1 month) to support treatment. On the first day after umbilical cord blood transfusion, the proportion of NK cells in peripheral blood are detected. If it is less than 20%, the NK cells are activated by subcutaneous injection of recombinant human interleukin-2 (rhIL-2) on the second day after infusion. The treatment effects are continuously monitored and followed up regularly after treatment.The intend of this trial is to explore whether cord blood transfusion in the consolidation phase can further reduce the recurrence rate of AML and improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Patients with primary AML diagnosed in accordance with the "Adult Acute Myeloid Leukemia (Non-Acute Promyelocytic Leukemia) Chinese Diagnosis and Treatment Guidelines (2017 Edition)", who achieved CR after induction chemotherapy
* Normal heart function , Ejection fraction ≥ 50%
* Normal liver function with ALT and AST ≤ 2.5 times the upper limit of normal value, bilirubin ≤ 2 times the upper limit of normal value
* Normal kidney function with blood creatinine ≤ 3.0 mg/dL (≤ 260 µmol/L)
* Voluntarily signed an informed consent.

Exclusion Criteria:

* Combined with severe infection
* Combined with other malignant tumors
* Other patients deemed unsuitable to be tested by the investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year Overall survival | 2-years
  the overall survival rate of enrolled patients at the end of 2 years

SECONDARY OUTCOMES:
2-year Disease-free survival | 2-years
  DFS is measured from the date when CR is achieved. And the end includes death or relapse.

CONTACTS AND LOCATIONS:
Overall Officials: huaiyu Wang, doctor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - The first affiliated hospital of Xi'an jiaotong university, Xi’an, Shanxi
  - Xi'anJiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
No sharing plan

REFERENCES:
- [Result] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Result] Li X, Dong Y, Li Y, Ren R, Wu W, Zhu H, Zhang Y, Hu J, Li J. Low-dose decitabine priming with intermediate-dose cytarabine followed by umbilical cord blood infusion as consolidation therapy for elderly patients with acute myeloid leukemia: a phase II single-arm study. BMC Cancer. 2019 Aug 20;19(1):819. doi: 10.1186/s12885-019-5975-8. PMID 31429724
- [Result] Dolstra H, Roeven MWH, Spanholtz J, Hangalapura BN, Tordoir M, Maas F, Leenders M, Bohme F, Kok N, Trilsbeek C, Paardekooper J, van der Waart AB, Westerweel PE, Snijders TJF, Cornelissen J, Bos G, Pruijt HFM, de Graaf AO, van der Reijden BA, Jansen JH, van der Meer A, Huls G, Cany J, Preijers F, Blijlevens NMA, Schaap NM. Successful Transfer of Umbilical Cord Blood CD34+ Hematopoietic Stem and Progenitor-derived NK Cells in Older Acute Myeloid Leukemia Patients. Clin Cancer Res. 2017 Aug 1;23(15):4107-4118. doi: 10.1158/1078-0432.CCR-16-2981. Epub 2017 Mar 9. PMID 28280089
- [Result] Ballen KK, Gluckman E, Broxmeyer HE. Umbilical cord blood transplantation: the first 25 years and beyond. Blood. 2013 Jul 25;122(4):491-8. doi: 10.1182/blood-2013-02-453175. Epub 2013 May 14. PMID 23673863
- [Result] Stringaris K, Sekine T, Khoder A, Alsuliman A, Razzaghi B, Sargeant R, Pavlu J, Brisley G, de Lavallade H, Sarvaria A, Marin D, Mielke S, Apperley JF, Shpall EJ, Barrett AJ, Rezvani K. Leukemia-induced phenotypic and functional defects in natural killer cells predict failure to achieve remission in acute myeloid leukemia. Haematologica. 2014 May;99(5):836-47. doi: 10.3324/haematol.2013.087536. Epub 2014 Jan 31. PMID 24488563
- [Result] Mehta RS, Shpall EJ, Rezvani K. Cord Blood as a Source of Natural Killer Cells. Front Med (Lausanne). 2016 Jan 5;2:93. doi: 10.3389/fmed.2015.00093. eCollection 2015. PMID 26779484